CLINICAL TRIAL: NCT06513013
Title: Comparative Evaluation of Magnesium Sulphate Versus Neostigmine as an Adjuvant to Bupivacaine in Ultrasound Guided Transversus Abdominis Plane (TAP) Block as Postoperative Analgesia in Cesarean Section
Brief Title: MgSO4 as Adjuvants to Bupivacaine vs Neostigmine in TAP Block in Cesarean Section
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alfarouk Ayman Farouk Omar, resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAP in cs using us
Record Dates: First submitted 2024-07-04; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Cesarean Section
Keywords: TAP; mg sulphate
MeSH Terms: interventions — Dental Occlusion; Cesarean Section; Magnesium Sulfate; Neostigmine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M "bupivacaine + normal saline + MgSO4" (Active Comparator): will receive 25 ml volume on each side ( 20 ml of 0.25% bupivacaine plus 5 ml of normal saline containing 250 mg of MgSO4 )
  Interventions: Procedure: transversus abdominis plane (TAP) block in cesarean section; Drug: Magnesium sulfate
- Group D "bupivacaine + normal saline + Neostigmine" (Active Comparator): will receive 25 ml volume on each side ( 20 ml of 0.25% bupivacaine plus 5 ml of normal saline containing 500 mcg of Neostigmine
  Interventions: Procedure: transversus abdominis plane (TAP) block in cesarean section; Drug: Neostigmine

INTERVENTIONS:
Procedure: transversus abdominis plane (TAP) block in cesarean section — .an intravenous (IV) access will be secured . Standard ASA monitoring will be instituted which include(SpO2), ECG and (NIBP) . At the end of surgery , a bilateral USG-guided TAP block will be carried out under strict aseptic precautions, and 20 mL of study solution was injected into each side. After draping the abdominal region between the 12th rib and anterior superior iliac crest with the umbilicus in the center, the external oblique muscle, internal oblique muscle, transversus abdominis muscle , and their fascia will be located beneath the skin and subcutaneous tissue using a linear high-frequency probe 6-13 Megahertz of the SonoSite Micromax machine. A 22-gauge spinal needle will be advanced using the in-plane technique at the anterior axillary line, and the precise position of the needle tip between the internal oblique and transverse abdominis muscle will be visualized. To expand the plane, 2 mL of normal saline will be administered.
Drug: Magnesium sulfate — 25ml volume on each side (20ml of 0.25% bupivacaine plus 5ml of normal saline containing 250 mg of MgSO4) to keep the total volume the same in both group
  Arms: Group M "bupivacaine + normal saline + MgSO4"
Drug: Neostigmine — 25ml volume on each side (20ml of 0.25% bupivacaine plus 5ml of normal saline containing 500 mcg neostigmine.
  A 22-gauge spinal needle will be advanced using the in-plane technique at the anterior axillary line, and the precise position of the needle tip between the internal oblique and transverse abdominis muscle will be visualized. To expand the plane, 2 mL of normal saline will be administered. Following the affirmation of a hypoechoic region on the USG image, the study solutions will be injected as per group allocation. Postoperatively,both groups of patients received an injection of paracetamol 1gm intravenously every 8th hourly as a part of multimodal analgesia and the patients will be evaluated for pain, nausea or vomiting in the post anaesthesia care unit at time 0 (time of completion of TAP block), 2, 4, 6,12 and 24 h by an investigator blinded to the group assignment. Whenever the NRS >4, Nalbuphine 0.1 mg/kg IV will be administered as a rescue analgesic.
  Arms: Group D "bupivacaine + normal saline + Neostigmine"

SUMMARY:
The aim of this study is to compare the duration of analgesia obtained by addition of Neostigmine versus MgSO4 as adjuvants to bupivacaine in TAP block in patients undergoing Cesarean Section and to evaluate postoperative analgesic requirements, side effects and level of patient satisfaction.

DETAILED DESCRIPTION:
Caesarean section (CS) is one of the most operations in the world. Effective postoperative analgesia after it is very important because it encourages breast feeding and facilitates early ambulation and recovery. Postoperative analgesia is too important to prevent unwanted side effects such as venous thromboembolism, respiratory complications and increased hospital stay.Post Caesarean discomfort and pain is expected; so, the analgesic regimen should assure safe and efficient sedation. Commonly, opioids and NSAIDs are used for post caesarean pain relief. While dose dependent respiratory depression is the most discomforting side effect, other insignificant side effects such as gastrointestinal upset, pruritus and urinary retention can be annoying during the first hours of puerperium. The transversus abdominus plane (TAP) block has been used for postoperative pain relief in different abdominal surgeries as part of the multimodal anesthetic approach.It creates satisfactory somatic anesthesia with no visceral blockade. Its widespread use in abdominal surgeries is due to its technical simplicity and trustworthy analgesia .This block implies administering local anesthetic between the internal oblique muscle and transversus abdominis muscle, which is marked by the lumbar Petit triangle. The primary drawback of single-shot regional blocks is their short duration of action when administered with local anesthetic alone. Several adjuvants, including opioids, alpha 2 agonists,Neostigmine, N-methylD-aspartate (NMDA) receptor antagonists, and other drugs, have been utilized to extend the duration of blocks . Opioids are by far the most often used adjuvants, but they accompany a host of unpleasant side effects, such as respiratory depression, drowsiness, nausea, and vomiting. In some studies, using alpha 2 agonists such as Dexmedetomidine and Clonidine has been related to drowsiness and bradycardia .

MgSO4 is an N-methyl-D-aspartate (NMDA) receptor antagonist. It acts by non-competitive antagonism blocking the voltage-dependent ion channels.

The potential of neostigmine as an adjuvant in peripheral nerve block is through its action to increase acetylcholine at muscarinic junctions of peripheral nerves. 500 mcg neostigmine was used as adjuvant to local anesthetic in an axillary brachial plexus block leads to decreased pain and less use of analgesics in the first 24 hours postoperatively with no incidence of adverse effects

ELIGIBILITY:
Inclusion Criteria:

* Age from 19 to 40 years old
* Singleton pregnencies with a gestational age of at least 37 weeks
* American society of anesthesiologists (ASA) physical state I , II
* patients undergoing spinal anesthesia for cesarean delivery via Pfannenstiel incision with exteriorization of the uterus.

Exclusion Criteria:

* Patient's refusal
* Age < 19 or > 40 years
* Height<150 cm, weight < 60 kg, body mass index (BMI) ≥40 kg/m2.
* Contraindications to spinal anesthesia (Coagulopathy, increased intracranial pressure, or local skin infection).
* Cardio-respiratory conditions
* Convulsions
* Inability to comprehend or participate in the pain scoring system.
* Bleeding diathesis
* Known allergy to any drugs used in this study

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-07-20 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
comparasion of Postoperative NRS score for 24 hours between the two groups | 24 hours postoperative
  NRS Score: used to assess pain intensity (13). It is one of the most commonly used pain scales in medicine. The NRS consists of a numeric version of the visual analog scale. It is a horizontal line with an eleven point numeric range. It is labeled from zero to ten, with zero being an example of someone with no pain and ten being the worst pain possible (Figure 2). This scale can be administered verbally. Rescue analgesia will be nalbuphine 0.1 mg/kg IV when the NRS ≥ 4.

SECONDARY OUTCOMES:
postoperative hemodynamic parameters | 24 hours postoperative
  Hemodynamic parameters including HR
time required for the first rescue analgesia | 24 hours postoperative
  the time at wich the patient demand analgesia will be record for each patient
total amount of rescue analgesic consumption duringfirst 24 hours postoperatively | 24 hours postoperative
  total amount of rescue analgesic consumption duringfirst 24 hours postoperatively
patient satisfacation score | 24 hours postoperative
  five-point likert scale: to evaluate the patient satisfacation regarding the
  to evaluate the patients' satisfaction regarding the whole procedure at the end of the postoperative 24 hours. It ranged from (1=very satisfied, 2=satisfied, 3=neither satisfied nor dissatisfied, 4=dissatisfied, 5=very dissatisfied)
PONV intensity by postoperatively: | 24 hours postoperative
  The number of attacks of nausea for 24 h will be assessed at 0.5, 1, 2, 4, 6, 12 and 24 h and will be recorded as yes/no.
  * The number of attacks of vomiting for 24 h will be assessed at 0.5, 1, 2, 4, 6, 12 and 24 h postoperatively and will be recorded as yes/no.

CONTACTS AND LOCATIONS:
Overall Officials: Zain Alabdin Zaree Hassan, Study Chair — Assiut University; Nashwa Farouk Abdel Hafez, Study Director — Assiut University

REFERENCES:
- [Background] Kapral S, Gollmann G, Waltl B, Likar R, Sladen RN, Weinstabl C, Lehofer F. Tramadol added to mepivacaine prolongs the duration of an axillary brachial plexus blockade. Anesth Analg. 1999 Apr;88(4):853-6. doi: 10.1097/00000539-199904000-00032. PMID 10195537
- [Background] Verma K, Malawat A, Jethava D, Jethava DD. Comparison of transversus abdominis plane block and quadratus lumborum block for post-caesarean section analgesia: A randomised clinical trial. Indian J Anaesth. 2019 Oct;63(10):820-826. doi: 10.4103/ija.IJA_61_19. Epub 2019 Oct 10. PMID 31649394
- [Background] Abrahams MS, Horn JL, Noles LM, Aziz MF. Evidence-based medicine: ultrasound guidance for truncal blocks. Reg Anesth Pain Med. 2010 Mar-Apr;35(2 Suppl):S36-42. doi: 10.1097/AAP.0b013e3181d32841. PMID 20216023